CLINICAL TRIAL: NCT00794144
Title: Safety and Pharmacokinetics of Patanase in Pediatric Patients 2 to < 6 Years of Age
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Cynthia M. Rusk\Manager, Development, Alcon Research
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: C-07-02
Record Dates: First submitted 2008-11-17; First posted 2008-11-19 (Estimated); Results first posted 2010-02-04 (Estimated); Last update posted 2010-03-04 (Estimated); Status verified 2010-02

CONDITIONS: Allergic Rhinitis
Keywords: Allergic Rhinitis; Pediatric; PATANASE
MeSH Terms: conditions — Rhinitis, Allergic

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Olopatadine Hydrochloride Nasal Spray 0.6%
  Interventions: Drug: Olopatadine Hydrochloride Nasal Spray 0.6%
- 2 (Placebo Comparator): Olopatadine Hydrochloride Nasal Spray Vehicle
  Interventions: Drug: Olopatadine Hydrochloride Nasal Spray Vehicle

INTERVENTIONS:
Drug: Olopatadine Hydrochloride Nasal Spray 0.6% — one spray in each nostril twice daily for 2 weeks
  Arms: 1
Drug: Olopatadine Hydrochloride Nasal Spray Vehicle — one spray in each nostril twice daily for 2 weeks
  Arms: 2

SUMMARY:
The purpose of the study is to assess the safety of the study drug, Patanase (Olopatadine Hydrochloride Nasal Spray 0.6%) compared to placebo (inactive substance) in children ages 2 to less than 6 who have a history of nasal allergies, and to assess the pharmcokinetics (study of the action of a drug in the body) in these children

ELIGIBILITY:
Inclusion Criteria:

* Patient must be at least 2 years of age and less than 6 years of age on Day 1;
* Parent/legal guardian must be willing and able to give written informed consent and must provide this consent for the study;
* Patient must have a positive case history of allergic rhinitis symptoms and at least one documented positive skin test within the 5 years prior to Day 1 of the following type: skin prick test, intradermal test or RAST test(radioallergosorbent test) for an allergen (≥ 3 mm wheal greater than diluent after skin prick testing; ≥ 7 mm wheal greater than the diluent after intradermal testing; or positive level 2 or greater after RAST testing);
* Patient and parent/caregiver must be willing and able to make required study visits;
* Patient and parent/caregiver must be able to follow instructions;
* Nasal exam must confirm absence of significant anatomic abnormalities, infection, bleeding, and mucosal ulcerations at Screening and prior to administration of test article at the Day 1 Visit. A finding of 'present' for any of these parameters disqualifies the patient from the study, regardless of clinical relevance.

Exclusion Criteria:

* The need for chronic or intermittent use of any prescription or over-the-counter nasal spray during the study period;
* Use of any form of olopatadine (e.g., PATANOL®, PATADAY™, PATANASE®) within 7 days of Day 1;
* Current or recent (within the last 14 days) use of any drugs/drug classes or combinations thereof that may prolong the QT interval;
* Patients with a history or evidence of nasolacrimal drainage system malfunction or abnormality that may interfere with the results of the study;
* Concurrent disease that might complicate or interfere with the investigation or evaluation of the study medications (such as rhinitis medicamentosa or large obstructive nasal polyps);
* Patients with syndromes associated with midfacial deformities or other anatomic nasal deformity that may interfere with the patient's participation in the study, as identified by physical or nasal examination at Screening or Day 1;
* Diagnosis of acute sinusitis within 30 days of Day 1 or diagnosis of chronic rhinosinusitis within one year of Day 1;
* Congestion that would, in the opinion of the investigator, interfere with successful nasal drug administration/absorption (in either nostril);
* Upper or lower respiratory infection within 14 days of Day 1;
* Asthma, with the exception of intermittent asthma as outlined in Section 18.5, from the Stepwise Approach for Managing Asthma in Children 0-4 Years of Age, and Stepwise Approach for Managing Asthma in Children 5-11 Years of Age (5);
* Current or recent (< 6 months) history of severe, unstable, or uncontrolled neurological, cardiovascular, gastrointestinal, hematological, hepatic, and/or renal disease, or evidence of other diseases at the physical examination conducted at the Screening Visit, which in the opinion of the Investigator would preclude the safe participation of the patient in the study;
* Hypersensitivity to olopatadine, benzalkonium chloride, or any component of the test articles;
* History or current infection of HIV (Human Immunodeficiency Virus), hepatitis B or C or A, as indicated by the patient's parent or legal guardian response on the HIV/Hepatitis survey;
* Relatives of study site staff or other individuals who would have access to the clinical study protocol;
* A family member or any individual residing in the same household of a patient that is currently enrolled in the study;
* Participation in any other investigational study within 30 days before entry into this study (Day 1), or concomitantly with this study;
* Clinically relevant abnormal vital signs (pulse rate, average systolic and diastolic blood pressure) at Screening or Day 1. The ranges below have been designated as normal for the study. Inclusion of patients with values outside of these normal ranges is at the discretion of the study investigator;

Normal Cardiovascular Ranges

* Systolic Blood Pressure - 86 to 116 mmHg (millimeters mercury)
* Diastolic Blood Pressure -50 to 78 mmHg
* Pulse - 75 to 130 bpm (beats per minute)

In addition, the Alcon Medical Monitor and/or Principal Investigator may declare any patient ineligible for the study based upon sound medical reasons.

Ages: 2 Years to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 132 (Actual)
Dates: Start 2008-10; Primary Completion 2008-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Niran Amar, MD, Principal Investigator; Sheri Byrd, MD, Principal Investigator — Spartanburg Medical Center; Albert Finn, MD, Principal Investigator — National Allergy, Asthma, & Urticaria; Joseph Flanagan, MD, Principal Investigator — Health Sciences Research Center; Brad H Goodman, MD, Principal Investigator — Aeroallergy Research Laboratories; Frank Hampel, MD, Principal Investigator — Central Texas Allergy and Asthma; Yu-Luen Hsu, MD, Principal Investigator — West Coast Clinical Trials Phase 2-4; Neil Kao, MD, Principal Investigator — Allergic Disease and Asthma Cente; John Prestigiacomo, MD, Principal Investigator — Gulf Coast Research Associates, Inc; Paul Ratner, MD, Principal Investigator — Sylvana Research Associates; Christopher Smith, MD, Principal Investigator — Asthma and Allergy Associates, P.C.
Locations (1):
- Niran Amar, M.D., Waco, Texas, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients at medical clinics in the U.S. participated from October 03, 2008, through December 03, 2008.
Pre-assignment Details: negative allergic response; enrollment target met
Groups:
- Olopatadine Hydrochloride Nasal Spray 0.6%: Olopatadine Hydrochloride Nasal Spray 0.6%
- Olopatadine Hydrochloride Nasal Spray Vehicle: Olopatadine Hydrochloride Nasal Spray Vehicle
Period: Overall Study
Arm/Group | Olopatadine Hydrochloride Nasal Spray 0.6% | Olopatadine Hydrochloride Nasal Spray Vehicle
Started | 66 | 66
Completed | 63 | 63
Not Completed | 3 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Olopatadine Hydrochloride Nasal Spray 0.6% | Olopatadine Hydrochloride Nasal Spray Vehicle | Total
Number analyzed (Participants) | 66 | 66 | 132
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 66 | 66 | 132
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28 | 36 | 64
  Male | 38 | 30 | 68

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Anatomic Nasal Exam Abnormalities
Description: The appearance in a participant of any of the following from Baseline: anatomic abnormalities, evidence of infection, bleeding, and/or ulcerations of the mucosa
Time Frame: Day 1 (Baseline) to Exit
Measure: Number; unit: Participants
Arm/Group | Olopatadine Hydrochloride Nasal Spray 0.6% | Olopatadine Hydrochloride Nasal Spray Vehicle
Number analyzed (Participants) | 66 | 66
Participants | 3 | 2

ADVERSE EVENTS:
Time Frame: 2 Weeks (Day 1 to Exit)
Description: Adverse events volunteered and solicited
Arm/Group | Olopatadine Hydrochloride Nasal Spray 0.6% | Olopatadine Hydrochloride Nasal Spray Vehicle
Serious Adverse Events (participants affected / at risk) | 0/66 | 0/66
Other Adverse Events (participants affected / at risk) | 15/66 | 14/66
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Olopatadine Hydrochloride Nasal Spray 0.6% (N=66) | Olopatadine Hydrochloride Nasal Spray Vehicle (N=66)
Cough (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 7 (7)
Pyrexia (General disorders) | 2 (2) | 6 (7)
Vomiting (Gastrointestinal disorders) | 3 (3) | 4 (4)
Diarrhoea (Gastrointestinal disorders) | 6 (6) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 1 (1)
Injury (Injury, poisoning and procedural complications) | 0 (0) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor reserves the right of prior review of any publication or presentation of information related to the study.